CLINICAL TRIAL: NCT01950754
Title: Study of the Effect of a Cognitive Task on Static Balance in Depressive Elderly Subjects According to the Double Task Principle
Acronym: DOUBLE TACHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: MANCKOUNDIA PHRC IR 2007
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Standing Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- depressive patients (Other)
  Interventions: Behavioral: standing with both feet; Behavioral: descent of the platform; Behavioral: standing on the platform, feet together and always with simultaneous performance of a task of mental count
- nondepressed controls (Other)
  Interventions: Behavioral: standing with both feet; Behavioral: descent of the platform; Behavioral: standing on the platform, feet together and always with simultaneous performance of a task of mental count

INTERVENTIONS:
Behavioral: standing with both feet
Behavioral: descent of the platform
Behavioral: standing on the platform, feet together and always with simultaneous performance of a task of mental count

SUMMARY:
This study could contribute to understanding the aggravation of balance disorders and the increased risk of falling in depressive people. It could, among other things, shed light on the impact of treatments with antidepressants on balance in treated depressive patients. Finally, it could contribute to improving the sensory-motor management of patients with a depressive syndrome.

ELIGIBILITY:
Inclusion Criteria:

In the 2 groups:

* General and cognitive status allowing the patient, according to the evaluation of the investigators, to take part in the study.
* Patients who provide written informed consent
* Patients covered by the national health insurance agency

In the "depression " group:

* Age ≥ 75 years,
* Subjects with a depressive syndrome, according to Geriatric Depression Scale criteria.
* Patients without treatment with antidepressants

In the "control" group:

* Age ≥ 75 years,
* Absence of a depressive syndrome

Exclusion Criteria:

In the 2 groups:

* Presence of a disabling orthopedic disease,
* Presence of any chronic neurological disease (cerebrovascular accident, Parkinson's syndrome …),
* Presence of a psychiatric disease apart from depression in the " depression " group
* Presence of a vestibular disease with clinical manifestations,
* Presence of a non-corrected visual disorder,
* Existence of a progressive organ disease,
* Psychotropic treatment able to impair vigilance and posture,
* Notion of one or several falls in the preceding 6 months,
* Oppositional personality or low motivation,
* Emotional or intellectual disorder.
* Patients under guardianship
* Patients who have taken part in a therapeutic trial in the previous 30 days

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-05-20 (Actual); Primary Completion 2013-05-14 (Actual)

PRIMARY OUTCOMES:
the difference in distance traveled by moving the center of pressure between the simple task and the dual task | up to 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France